CLINICAL TRIAL: NCT00301613
Title: MMF Versus Intravenous CTX Pulses in the Treatment of Adult Severe Henoch-Schonlein Purpura Nephritis
Brief Title: Mycophenolate Mofetil (MMF) Versus Intravenous CTX Pulses in the Treatment of Adult Severe HSPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0605
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2008-07

CONDITIONS: Henoch-Schoenlein Purpura; Nephritis
Keywords: Henoch-Schonlein purpura nephritis Mycophenolate mofetil; Cyclophosphamide; treatment
MeSH Terms: conditions — IgA Vasculitis; Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mycophenolate mofetil (Active Comparator)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — MMF,1.0g/d
  Other Names: Mycophenolate mofetil,cellcept

SUMMARY:
This study is performed to compare the efficacy, safety, tolerability and relapse of MMF vs CTX in the treatment of severe HSPN

DETAILED DESCRIPTION:
Henoch-Schoenlein purpura nephritis (HSPN) with massive proteinuria,renal insufficiency and crescent formation at onset have high risks of progressing to end stage renal failure. Though clinical studies have shown that steroids in combination with cyclophosphamide could reduce proteinuria and preserve renal function, this protocol is associated with many side effects, and is not effective in some patients.

Recent studies have shown that mycophenolic acid(MPA), the active metabolite of mycophenolate mofetil(MMF),could inhibit multifarious effects on endothelial cells, including adhesion molecular expression, neutrophil attachment,IL-6 secretion, and the process of angiogenesis, which contribute to the efficacy of MMF in the treatment of vasculitis. Clinical studies also showed that MMF was effective in the treatment of lupus nephritis with vasculitic lesions. These findings suggest that MMF might be effective in the treatment of severe HSPN, which is a kind of vasculitic lesion. This prospective open-labeled clinical trial study investigates the efficiency of MMF in the treatment of severe HSPN compared with pulse intravenous cyclophosphamide. After 12 months of treatment, we will assess the efficacy, safety, tolerability and relapse of MMF compared with cyclophosphamide in the treatment of severe HSPN.

ELIGIBILITY:
Inclusion Criteria:

* 16-50 years
* Biopsy proved HSP
* Proteinuria ≥ 3.0 g/24hr
* Scr < 5.0 mg/dl

Exclusion Criteria:

* Cytotoxic drug treatment such as CTX, CsA, MMF for morn than 1 month-3 months prior to enrolled
* Pregnancy
* Active/serious infections
* Previous diagnosed diabetes mellitus type 1 or 2

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2003-01; Primary Completion 2005-05 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy,safety, tolerability and relapse of MMF vs CTX in the treatment of severe HSPN | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hong Liu, M.D., Study Chair — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224